CLINICAL TRIAL: NCT07194395
Title: A Prospective International Multicenter, Non-Interventional, Single Arm, Blinded Feasibility Study to Assess the Contactless Optical Monitoring of AV Access Using the PatenSee System in Dialysis Patients
Brief Title: Contactless Optical Monitoring of AV Access Using the PatenSee System in Outpatient Hemodialysis Patients
Status: Recruiting | Type: Observational
Sponsor: PatenSee Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CMAP-001
Record Dates: First submitted 2025-09-10; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Hemodialysis; Clinical Assessment
Keywords: Nephrology; AV access; Clinical monitoring of AV access; Fistula; AV graft
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AVF/G access: Patients with AV access (AVF/G) undergoing hemodialysis
  Interventions: Device: PatenSee System

INTERVENTIONS:
Device: PatenSee System — Contactless AV access monitoring device

SUMMARY:
This is a prospective, non-interventional, single arm, international multicenter study in which up to 120 adult participants with kidney failure requiring regular hemodialysis through arteriovenous (AV) access (AV fistula or graft) will be recruited and evaluated using the PatenSee system.

Data captured on the PatenSee system will be analyzed and evaluated against standard of care clinical monitoring of AV accesses.

DETAILED DESCRIPTION:
For eligible participants, a clinical exam of the AV access ("Look, Listen, Feel") per SOC will be done by a qualified site clinician/nurse, followed by an assessment of the AV access using the PatenSee system on a weekly basis for 6 weeks, and then biweekly up to 1 year from enrollment. Additional data regarding imaging and complications of the AV access will be collected. Clinical decisions, such as referrals for further investigation and management of the AV access will be based solely on standard clinical monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult patient aged ≥18 years old
2. Patient has a non-reversible kidney failure that requires long-term hemodialysis
3. Patient has a functioning AV access (AVF/G) in the upper extremity
4. Patient is able and willing to provide consent by signing an EC/IRB approved informed consent form
5. Patient is willing and able to follow the requirements of the study

Exclusion Criteria:

1. An active AV access infection
2. An AV access condition that will likely require revision, e.g., symptomatic steal syndrome
3. Expected to recover kidney function, receive a kidney transplant, transfer to peritoneal dialysis (PD) or transfer to non-study site during the study period.
4. Any reason per investigator's discretion for which the patient is not suitable for the study
5. Any medical or psychiatric illness, which in the opinion of the investigator would compromise the patient's ability to adhere to study requirements
6. Previous participation in an interventional study within 30 days prior to study enrollment that may interfere with evaluation of the study endpoints
7. Female patient is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary dialysis clinics
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Comparison of "Look" assessment with PatenSee's relevant output | 6 weeks per patient
  Agreement between the ability to detect AV access structure parameters by PatenSee's images and the ability to detect the same parameters by clinical monitoring
Comparison of "Listen & Feel" assessments with PatenSee's relevant output | 6 weeks per patient
  Agreement between the PatenSee audio analysis of the AV access bruit and the sound recording of the AV access using a standard digital stethoscope measured

SECONDARY OUTCOMES:
Functionality endpoint - Average time to conduct PatenSee scanning data capture | Up to 12 months
  Average time to conduct PatenSee scanning data capture
Functionality endpoint - Proportion (%) of participants on whom the PatenSee was used as planned | Up to 12 months
  Proportion (%) of participants on whom the PatenSee was used as planned
Functionality endpoint - Average number of weeks participants obtained PatenSee measurements | Up to 12 months
  Average number of weeks participants obtained PatenSee measurements

OTHER OUTCOMES:
Safety Endpoints - Assessment of device related AEs | Up to 12 months
  Assessment of device related AEs
Exploratory Endpoints - AV access data collection | Up to 12 months
  Data collected in the study will be used to train PatenSee system's ability to alert on stenosis and other signs of AV access dysfunction processes.

CONTACTS AND LOCATIONS:
Locations (2):
- Henry Ford Hospital, Detroit, Michigan, United States
- Meir Medical Center, Kfar Saba, Hasharon, Israel

IPD SHARING:
Plan to Share IPD: No